CLINICAL TRIAL: NCT00464841
Title: Can the Tsui Test be Used to Test the Placement of Epidural Catheters Following the Intrathecal Component of a Combined Spinal-epidural Technique Used for Labor Analgesia?
Brief Title: Usefulness of the Tsui Test in Combined Spinal-Epidural Analgesia in Labour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-02; 06-0205-A
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Labor Pain
Keywords: Tsui Test; Combined Spinal Epidural; Labour
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Tsui test for combined spinal-epidural
  Interventions: Procedure: Combined spinal epidural
- 2 (Experimental): Tsui test for intrathecal catheter
  Interventions: Procedure: Tsui Test for intrathecal catheter

INTERVENTIONS:
Procedure: Combined spinal epidural — 0.7 mL of 0.25% isobaric bupivacaine and 15mcg of fentanyl
  Arms: 1
Procedure: Tsui Test for intrathecal catheter — 0.7 mL of 0.25% isobaric bupivacaine and 15mcg of fentanyl
  Arms: 2

SUMMARY:
Combined spinal epidural anesthesia (CSE) is a very effective technique to provide labor analgesia. One of the disadvantages of this technique is the delay in recognizing an error in the position of the epidural catheter because of the effects of the spinal component. Eventually in case of a misplaced catheter, the patient will experience pain or discomfort requiring a repeat procedure after the effect of drug given during the spinal wears off. Low current electrical stimulation test, or the Tsui test, has been used successfully to confirm catheter location in the epidural space. The investigators' objective in this study is to test the usefulness of the Tsui test to confirm the correct placement of the epidural catheter during CSE in laboring patients.

DETAILED DESCRIPTION:
CSE is a widely used technique to provide analgesia in laboring patients. One of the disadvantages of the CSE is the delay in recognizing the mal-position of the epidural catheter, which is initially masked due to the effects of the spinal component. A mal-positioned epidural catheter can cause unnecessary maternal discomfort and dissatisfaction, as it requires a repeat procedure when the effect of spinal drug wears off. Additionally, in the event of emergency caesarean delivery, it would be advantageous to know that the catheter is properly placed. Low current electrical stimulation test, or the Tsui test, has been used successfully to confirm catheter location in the epidural space. Our objective in this study is to test the usefulness of the Tsui test to confirm the correct placement of the epidural catheter during CSE in laboring patients.

Two groups of patients will be studied. In the first group, after the placement of the epidural catheter and noting the electric current required to elicit a motor response (maximum current used is 20 mA), a spinal needle is introduced one inter vertebral space below the space where the epidural catheter is inserted and 0.7 ml of 0.25% isobaric bupivacaine and 15 mcg of fentanyl is injected intrathecally. The epidural catheter is then re-stimulated and the magnitude of the current required to reproduce the motor response is noted. The stimulation is repeated after 5, 10, and 15 minutes. The second group consists of patients with accidental dural puncture. An intrathecal catheter is inserted and the Tsui test performed (maximum current used is 2 mA), followed by the injection of same mixture of local anesthetic and opioid as used in the first group. The Tsui test is repeated at 5, 10 and 15 minute intervals, similar to what is done in the epidural group. After 15 minutes, patients in both groups are managed as per departmental policy. In both the groups, the Tsui test will be repeated after 120 minutes during the maintenance of labor analgesia to determine the change in intensity of current required to elicit the motor response.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) 1 or 2
* Full term pregnancy
* Patients requesting epidural in early labor

Exclusion Criteria:

* Any contraindication to regional anesthesia
* Allergy or hypersensitivity to lidocaine, bupivacaine, or fentanyl
* Received prior sedatives or opioids
* Abnormal vertebral anatomy
* Neurological disorders with lumbar involvement
* Patients with implanted electronic devices

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
change in current intensity required to produce a positive Tsui test after an intrathecal injection of bupivacaine | Within 2 hours of catheter placement

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, PhD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Carvalho JC, Khemka R, Loke J, Tsui BC. Low-dose intrathecal local anesthetic does not increase the threshold current for the epidural stimulation test: a prospective observational trial of neuraxial analgesia in labouring women. Can J Anaesth. 2015 Mar;62(3):265-70. doi: 10.1007/s12630-014-0291-x. Epub 2014 Dec 11. PMID 25501494